CLINICAL TRIAL: NCT04642248
Title: A Comprehensive Analysis for Identification of Risk Factors for Running-Related Injuries
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ACE Running LLC (Industry)
Collaborators: Air Force (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Pre-BMT Run
Record Dates: First submitted 2020-10-30; First posted 2020-11-24 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Runner's Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-intervention (Active Comparator): This group will have the analysis and their data will be used to determine risk factors for developing running injuries.
  Interventions: Other: Personalized Run Practice
- Intervention (Experimental): This group will get a personalized program based off of 3D and movement analysis results to judge the ability to reduce musculoskeletal injuries.
  Interventions: Other: Personalized Run Practice

INTERVENTIONS:
Other: Personalized Run Practice — A combination of drills, flexibility, and strength activities combined with a gait retraining program

SUMMARY:
At a basic level, running-related injuries (RRI) occur because the forces acting on the body exceed the capacity of the tissue to absorb the forces causing a breakdown of the tissue. When looking at ways to reduce RRI, the general strategy should be to make the body's ability to absorb forces greater than the forces acting on it. This can be accomplished by improving flexibility, increasing strength, reducing participation, improving recovery, and finally improving running form through gait retraining. Due to constraints of research by the ability to get large enough data sets, most literature has looked at one of these ways to make the forces manageable for a runner, while there are many ways. Running is not the only time that the body absorbs forces. This is especially true in a military population where there is a cumulative effect of forces from marching with heavy load, prolonged standing, and limited recovery.

Gait retraining has been shown to reduce injury rates by as much as 60%. Two studies have looked specifically at military populations to show that gait retraining can be effective for reducing a common injury in the shin. Military studies have also shown that gait retraining is transferable to wearing boots, even when the gait retraining is done in shoes. In the commercial sector, many studies have shown the benefit of changing running form with cadence modification, increasing forward lean, reducing collapsing at the knee, and modifying the position of the foot when the foot hits the ground. The aim of this study is taking the best evidence from gait retraining efforts and personalize the methodology to the individual runner. No study to date has provided individual recommendations for gait retraining, nor has the capabilities to do so that this portable 3D motion analysis system provides. The results can be used on a large scale to have a significant reduction in RRI and a monumental benefit to society.

DETAILED DESCRIPTION:
The total project will last 12 months, with 3 months to prepare testing facilities and train personnel, 6 months to analyze enough subjects for statistical power, and 3 months of statistical analysis and review. Between three to eleven Air Force Reserve bases with a Developmental Training Flight (DTF) will be given a RunDNA 3D Motion Analysis system to participate as testing facilities. The DTF is part of the Air Force Reserves where new recruits undergo education and training prior to BMT. Three to five Exercise Physiologists at each DTF base will be trained on how to perform the RunDNA analysis. Training will be done remotely, which has already successfully been done through video-based lectures at 6 Air Force bases. Each research examiner will pass a test and must submit a 3D analysis done with the RunDNA device prior to testing for standardization of procedures.

Each DTF has upwards of 100 military recruits who are preparing to attend BMT at any given time. Recruits will undergo baseline fitness testing when they are within 16 weeks of attending BMT. Fitness testing is comprised of a timed mile and a half run, two-minute timed pushup test, and two-minute timed sit up test. Three days or less after Fitness Testing (once any soreness has resolved), the recruits will undergo the RunDNA Analysis.

The RunDNA analysis consists of a Running Readiness Assessment (RRA) to determine mobility and strength and a 3D gait analysis to assess running form. The RRA is comprised of thirteen movement-based assessments that are scored with specific criteria for each test. The tests are:

1. Toe Touch
2. Back Bend
3. Rotation
4. Single Leg Balance - Eyes Closed
5. Squat
6. Single leg sit to stand
7. Unilateral Hip Bridge Endurance Test
8. Single Leg Calf Raise
9. Side Plank
10. Toe Splay
11. Hallux Extension
12. Hallux Abduction
13. Ankle Range of Motion Items 1 through 5 have additional break downs to further identify limitations in movement and prescribe specific corrective exercise programs. DTF site personnel will enter the RRA results into the RunDNA mobile app at the time of administration. A scoring system has been created for a total of 55 points, where 1 point is given for a strength limitation, 2 points for a mobility limitation, and 3 points for painful movement. Each runner will be given a score from their RRA.

The 3D running analysis will use a portable device mounted on a tripod five feet behind a treadmill. There are 3 optical motion capture cameras with LED lights in each device. Eighteen reflective markers will be adhered to each runner using the modified Helen Hayes protocol. Runners will be given a minimum of 2 minutes to warm up, and then 15 seconds of running will be captured. After the quality of the 3D capture has been verified, each runner will be assigned a running category determined by the software. The software will communicate the running category with the mobile app and the groups that are being prescribed exercises will have those programs added to their profile.

Research participants (recruits) will also fill out information on demographics, running experience, and injury history under their profile in the mobile application.

Investigators will randomly assigning which participants will be getting the intervention program at the DTF sites to prescribe personalized programs based off the RunDNA analysis. Examiners will assign the program based off of the user id that is generate, where odds will be give the intervention and evens will not. The prescription of the programs is standardized by using the mobile app to analyze the runner's results and prescribe one corrective exercise program from the RRA, one gait category program, and one fitness training program. The gait category program will be one of twelve programs that classify runners after the software analyzes all running variables. Each category has specific warm up exercises, specific drills, and specific gait retraining methods to lower the risk of injury for runners by improving their form. An example category is an overstrider cadence program. This person lands with the foot too far in front of the body because they have a slow step rate. The overstrider cadence program includes a dynamic warm up, drills using a higher step rate, and gait retraining where the runner matches their footsteps to a metronome that is 5-10% higher than their self-selected step rate.

Recruits will go through a minimum of 8 weeks of training at DTF using the mobile app and GPS watches to track compliance and training loads. The training program utilizes motor learning principles to gradually increase the time a runner uses the new form with faded feedback to allow for a natural adoption of the running technique. Cross training is included for cardiovascular fitness, as well as speed work for running in the later stages of the program to improve performance. Within 2 weeks of the recruit going to BMT, site personnel will readminister the Fitness Tests and RunDNA Analysis using the same procedures listed above to monitor changes in fitness, mobility, strength, and running form. Results will be recorded in the RunDNA app for analysis.

All recruits will be monitored through the mobile application during BMT to assess Fitness Test performance, injury rates, utilization of medical services, graduation rate, and subjective pain and fatigue reports. Recruits will continue to wear the GPS device to track training load. A daily subjective questionnaire will be filled out by the recruits on their issued iPad reporting on injury status and syncing the watch's training data. If iPads are not available to use the RunDNA app for each recruit, an analogue journal will be provided that has their research subject number in the journal. Each recruit will be given their subject number to know which journal is theirs. At the end of BMT the journals will be mailed to be manually entered. If iPads are not available to use the RunDNA app, multiple iPads will be sent to the medical staff at BMT and participants will come in twice weekly to sync their GPS device with the iPad to load up training data from the GPS.

There will be no change in training plans from standard BMT protocols for recruits doing through this research study. If at any point a recruit experiences injury or requests medical attention the BMT medical staff will alert the Principle Investigator.

Statistical analysis will be done on all results to answer the primary research question, with the anticipation of identifying key modifiable variables related to running injuries in the control group and the intervention group's ability to reduce injury rates and boost performance.

ELIGIBILITY:
Inclusion Criteria:

* Attending Basic Military Training

Exclusion Criteria:

* No active or past injury within 6 months that precluded them from participating in physical activity or that they sought medical attention for; No medical profile that excludes them from running

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Running Related Injury | Up to 24 weeks from DTF to Completion of BMT
  A daily questionnaire will be filled out by participants. There are four questions that identify injury status, pain, perceived ability to perform at their best, and changes in daily activities that may relate to injury or performance. Participants that answer "no" to the Question: "Are you physically able to run today" will be assessed for injury status and this will be monitored during the study.

IPD SHARING:
Plan to Share IPD: No